CLINICAL TRIAL: NCT03041493
Title: Investigation of the Effects of Electronic Cigarettes on Vascular Health
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of accrual
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 17-071
Record Dates: First submitted 2017-02-01; First posted 2017-02-02 (Estimated); Last update posted 2021-06-18 (Actual); Status verified 2021-06

CONDITIONS: Vascular Health
Keywords: Electronic Cigarettes; 17-071
MeSH Terms: conditions — Vaping | interventions — Electronic Nicotine Delivery Systems

STUDY DESIGN:
Intervention Model Description: This is a prospective, non-randomized case controlled study of the effects of electronic cigarettes on vascular health. The study population will comprise the three groups based on the criteria EC users (experimental group), (TC) smokers (positive control) and nonsmokers (negative control).
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Electronic cigarettes (EC) smokers (Experimental)
  Interventions: Behavioral: Electronic cigarette
- traditional cigarette (TC) smokers (Experimental)
  Interventions: Behavioral: traditional cigarette
- nonsmokers (Active Comparator)
  Interventions: Behavioral: (sham cigarette) - no actual exposure to cigarettes

INTERVENTIONS:
Behavioral: Electronic cigarette — During the first encounter, blood pressure and endothelium-dependent relaxation (EDR) will be measured by flow mediated dilatation (FMD), and a small peripheral IV catheter will be placed in the participant's median antecubital or cephalic vein. A blood sample (10 mL) for EPCs and F2-isoprostanes will be collected. One urine sample will also be collected for measurement of urinary F2-isoprostanes, cotinine and creatinine. These will serve as both baseline measures for subsequent acute exposure to nicotine and as measures of chronic nicotine exposure. The second encounter will be scheduled 4 hours after the first encounter. At that time a blood sample (5 mL) for EPCs will be collected followed by harvesting of vascular endothelial cells for eNOS and NF-κB expression.
  Arms: Electronic cigarettes (EC) smokers
Behavioral: traditional cigarette — During the first encounter, blood pressure and endothelium-dependent relaxation (EDR) will be measured by flow mediated dilatation (FMD), and a small peripheral IV catheter will be placed in the participant's median antecubital or cephalic vein. A blood sample (10 mL) for EPCs and F2-isoprostanes will be collected. One urine sample will also be collected for measurement of urinary F2-isoprostanes, cotinine and creatinine. These will serve as both baseline measures for subsequent acute exposure to nicotine and as measures of chronic nicotine exposure. The second encounter will be scheduled 4 hours after the first encounter. At that time a blood sample (5 mL) for EPCs will be collected followed by harvesting of vascular endothelial cells for eNOS and NF-κB expression.
  Arms: traditional cigarette (TC) smokers
Behavioral: (sham cigarette) - no actual exposure to cigarettes — During the first encounter, blood pressure and endothelium-dependent relaxation (EDR) will be measured by flow mediated dilatation (FMD), and a small peripheral IV catheter will be placed in the participant's median antecubital or cephalic vein. A blood sample (10 mL) for EPCs and F2-isoprostanes will be collected. One urine sample will also be collected for measurement of urinary F2-isoprostanes, cotinine and creatinine. These will be compared to the second set of laboratory measurements done at the second encounter that will be scheduled 4 hours after the first encounter. At that time an additional blood sample (5 mL) for EPCs will be collected followed by harvesting of vascular endothelial cells for eNOS and NF-κB expression.
  Arms: nonsmokers

SUMMARY:
The goal is find out if the use of Electronic cigarettes (EC) leads to the same changes that we see in blood vessels of traditional cigarettes (TC) users. The investigators will also enroll non-smokers as "controls", against which they will measure changes in blood vessels in TC and EC users.

ELIGIBILITY:
Inclusion Criteria:

* Male or female between 18 and 50 years of age.
* Good general health with no history of diabetes, coronary artery disease, peripheral arterial disease, chronic disease or hypertension.
* Ability to sign an informed consent.

Tobacco product users will have additional inclusion criteria:

* For TC smokers, daily TC smoking in the past 6 months, at least 10 cigarettes per day, with no EC exposure in the past 6 months
* For EC users, daily EC use in the past 6 months, at least 10 sessions per day, with no TC exposure in the past 6 month
* For non-smokers, no significant lifetime exposure to any nicotine-containing product, where significant exposure is defined as daily use of any nicotine-containing product for more than one week or once monthly use for more than 6 months.

Exclusion Criteria:

* History of renal disease, hypertension, diabetes, congestive heart failure or emphysema
* Use of ACE inhibitors, Angiotensin II receptor blockers, diuretics, aldosterone, renin blockers, aspirin, statins, sildenafil (or other PDE5 inhibitors) and NSAIDs.
* History of substance abuse
* Currently using nicotine replacement or other tobacco cessation products or intentionally abstaining from nicotine-containing products
* IV contrast exposure in the past 1 month
* Inability to place an IV catheter or draw blood for any reason
* Pregnant women or breastfeeding

  * Potential subjects will be asked if they are pregnant. Verbal confirmation of pregnancy will be sufficient.
* Fever of >101°F or BP >180/95
* BMI ≥30

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2021-06-11 (Actual); Study Completion 2021-06-11 (Actual)

PRIMARY OUTCOMES:
Differences in levels of F2-isoprostanes in participants | 2 years
  F2-isoprostanes in blood and urine

CONTACTS AND LOCATIONS:
Overall Officials: Roman Shingarev, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm